CLINICAL TRIAL: NCT02589457
Title: A Randomized, Open-label, Single-dosing, 2x2 Crossover Study to Compare the Safety and Pharmacokinetics of CKD-390 Tablet (Tenofovir Disoproxil Aspartate) With Viread® Tablet (Tenofovir Disoproxil Fumarate) in Healthy Male Volunteers
Brief Title: Study to Compare the Safety and Pharmacokinetics of CKD-390 Tablet With Viread® Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 163BE15028
Record Dates: First submitted 2015-10-06; First posted 2015-10-28 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B virus, HIV-1 infection; Healthy Male Volunteer; Tenofovir Disoproxil Fumarate
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Viread® tablet (Active Comparator): Tenofovir Disoproxil Fumarate
  Interventions: Drug: Viread® tablet
- CKD-390 (Experimental): Tenofovir Disoproxil Fumarate
  Interventions: Drug: CKD-390

INTERVENTIONS:
Drug: CKD-390 — Tenofovir Disoproxil Aspartate 1T PO
  Arms: CKD-390
Drug: Viread® tablet — Tenofovir Disoproxil Fumarate 1T PO
  Arms: Viread® tablet

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetics of CKD-390(Tenofovir Disoproxil Aspartate) and Viread® tablet(Tenofovir Disoproxil Fumarate) in healthy male volunteers.

DETAILED DESCRIPTION:
A Randomized, Open-label, Single-dosing, 2x2 Crossover Study to Compare the Safety and Pharmacokinetics of CKD-390 Tablet (Tenofovir Disoproxil Aspartate) With Viread® Tablet (Tenofovir Disoproxil Fumarate) in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer in the age of 19-45
2. Body weight ≥ 55kg and in the range of calculated Ideal Body Weight ± 20%
3. Subject without a hereditary problems, chronic disease and morbid symptom
4. Subject who sign on an informed consent form willingly

Exclusion Criteria:

1. Clinically significant disease with hepatobiliary, nephrological, gastrointestinal, respiratory, hepato-oncological, endocrine, urogenital, neurologic, psychiatric, musculoskeletal, immune, otorhinolaryngological, cardiovascular system
2. Gastrointestinal disease(Crohn's disease, ulcer, acute/chronic pancreatitis) or gastrointestinal surgery(except for appendectomy or herniotomy)
3. Hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of drugs or additives
4. Galactose intolerance, Lapp lactase deficiency or Glucose-galactose malabsorption
5. Sitting systolic blood pressure > 140mmHg or < 100mmHg, sitting diastolic blood pressure ≥ 90mmHg or < 60mmHg, pulse ≥ 100 beats per minute
6. Aspartate aminotransferase, Alanine aminotransferase, Total bilirubin > 2 x upper limit of normal range
7. Have the result of Creatinine clearance is less than 50mL/min(Cockcroft-Gault equation applicable)
8. The history of drug abuse or drug abuse showed a positive for urine drug test
9. Subject treated metabolizing enzyme inducers or inhibitors including barbiturates within 1 month
10. Subject treated ethical the counter or herbal medicine within 2 weeks, over-the-counter or vitamin within 1 week
11. Taking drugs have received any other investigational drug within 3 months prior to the first dosing
12. Whole blood donation within 2 months prior to the first dosing or component blood donation within 1 months prior to the first dosing or blood transfusion within 1 month
13. Continuously taking excessive alcohol (> 21 units/week; 1 unit = 10g of pure alcohol) or cannot stop drinking from 24 hours before admission to discharge
14. Cigarette > 10 cigarettes a day on average for recent 3 months
15. Subjects with planning of dental treatment (tooth extraction, endodontic treatment etc.) and any surgery (aesthetic operation, laser in-situ keratomileusis, laser assisted sub-epithelial keratomileusis etc.) from signed on an informed consent form to post-study visit
16. An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
AUCt of Tenofovir | 0(Pre-dose) up to 72hr

SECONDARY OUTCOMES:
AUCinf | 0(Pre-dose) up to 72hr
Blood pressure | 1 day, 2 day, 3 day, 4 day, 15 day 16 day, 17 day 18 day, 25 day
tmax | 0(Pre-dose) up to 72hr
t1/2β | 0(Pre-dose) up to 72hr
Clearance/F | 0(Pre-dose) up to 72hr
Electrocardiography | 1 day, 2 day, 3 day, 4 day, 15 day 16 day, 17 day 18 day, 25 day
Physical Examination | 1 day, 2 day, 3 day, 4 day, 15 day 16 day, 17 day 18 day, 25 day
Pulse rate | 1 day, 2 day, 3 day, 4 day, 15 day 16 day, 17 day 18 day, 25 day
Temperature | 1 day, 2 day, 3 day, 4 day, 15 day 16 day, 17 day 18 day, 25 day

CONTACTS AND LOCATIONS:
Overall Officials: Jang Hee Hong, MD, PhD, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, Jung-gu, South Korea